CLINICAL TRIAL: NCT01199666
Title: Text 4 Health-Kids: Text Message Reminder-Recalls For Early Childhood Vaccination
Brief Title: Text Message Reminder-Recalls For Early Childhood Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Melissa Stockwell, MD, MPH, Asst Prof of Pediatrics and Population and Family Health, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AAAF4263
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Vaccination
Keywords: Underimmunization, text message, vaccination; Underimmunization

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text message reminders (Experimental)
  Interventions: Other: Text message
- standard of care for MMR, letter reminder for Hep A (Active Comparator): MMR: automated phone call appointment reminder Hep A: recall letter, automated phone call appointment reminder
  Interventions: Other: Text message

INTERVENTIONS:
Other: Text message — text message appointment and immunization reminders

SUMMARY:
Although the investigators have reached the Healthy People 2010 goal of 80% coverage among U.S. children 19-35 months of age for the primary immunization series, 20% of children still remain underimmunized. In addition, pockets of low immunization coverage and outbreaks of vaccine preventable disease persist. Immunization reminder-recalls have been shown to be successful, but have been limited by the ability to identify and reach large target populations in a real-time, automated fashion. Reminder-recalls via text message may offer an innovative opportunity to improve vaccination coverage. Currently, 91% of Americans own a cell phone. Prior research by our team suggests that text messages reminder recalls may be an effective tool to remind parents about their children's vaccines. In this study, the investigators will demonstrate the effectiveness of tailored text message appointment and immunization reminders linked to a well-established and functional immunization registry to increase coverage rates and timeliness of the sentinel vaccines of MMR and HepA. The investigators will target parents of young children from an underserved population that is primarily Latino, with low socioeconomic status.

ELIGIBILITY:
Inclusion Criteria:

* Parents of child >9 months to 25 months
* Child with at least one visit to one of the participating clinical sites in the previous 12 months
* Parental cell phone number recorded in the registration system

Ages: 9 Months to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2586 (Actual)
Dates: Start 2011-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Receipt of MMR1 | by 13 and 16 months of age

SECONDARY OUTCOMES:
Timeliness of HepA vaccination post-recall | 4,12, 24 weeks
Attendance at appointments | after appointment

CONTACTS AND LOCATIONS:
Overall Officials: Melissa S Stockwell, MD MPH, Principal Investigator — Columbia University; Annika Hofstetter, MD PhD MPH, Study Director — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States